CLINICAL TRIAL: NCT02007681
Title: The Effects of Shifting Sedentary Behaviors to Light Activities on Energy Expenditure: A Randomized Controlled Trial in Sedentary Adults
Brief Title: What is in Fact the Contribution of Reducing Time Spent in Sedentary Behaviors on Daily Energy Expenditure? A Doubly Labeled Water Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Lisbon (Other)
Responsible Party: Principal Investigator, Analiza M Silva, PhD, Analiza M Silva, Technical University of Lisbon
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CEFMH || Parecer 14/2013
Record Dates: First submitted 2013-11-26; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Risk Reduction Behavior
Keywords: Sedentary Behavior; Breaks; Workplace; Energy Expenditure; Physical activity; doubly labeled water
MeSH Terms: conditions — Risk Reduction Behavior; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle change (Experimental): One 5-10 minute break per hour during the work day using a software that alert the participant, and perform 6000 steps above the baseline number of steps/day (previously evaluated), by adopting several domain specific strategies, during 7 days.
  Interventions: Behavioral: Reduction of sedentary time by breaking it with low intensity physical activity
- Control (No Intervention): Regular free week with no changes performed

INTERVENTIONS:
Behavioral: Reduction of sedentary time by breaking it with low intensity physical activity — One 5-10 minute break per hour during the work day using a software that alert the participant, and perform 6000 steps above the baseline number of steps/day (previously evaluated), by adopting several domain specific strategies, during 7 days.
  Other Names: LIPA; breaks
  Arms: Lifestyle change

SUMMARY:
The main purposes of this randomized cross-over trial are to test if a 3h/day reduction of time spent in sedentary behaviour (SB) through breaking up hourly and shifting it for standing and walking behaviours would substantially increase total (TEE) and PA energy expenditure (PAEE) compared to a week of habitual prolonged SB, in male and female overweight/obese inactive (which do not attained MVPA recommendations) and sedentary desk workers. Specifically using an experiment design our main aims are: a) to determine the impact of reducing SB on TEE and PAEE; b) to analyse the independent effects of interrupting SB through breaks and the overall reduction in SB on TEE and PAEE; c) To analyse the determinants for the overall reduction in SB; d) If the changes occurred in TEE and PAEE were dependent on specific covariates.

DETAILED DESCRIPTION:
There is enough information about exercise physiology to support the well-documented public health guidelines promoting at least 150 minutes of moderate-to vigorous physical activity (MVPA)(1). However there is an emergence of inactivity physiology studies. If we divide a day into periods of MVPA, light intensity PA (LIPA), sedentary behavior and sleep we observe a large proportion of the time taken up by time spent sitting, such as TV viewing, car driving and computer use. In fact, evidence exists that excessive time spent in sedentary behavior (SB) is a health risk that is not mitigated by performing half an hour of MVPA per day (2, 3). Life expectancy at birth may increase by ~2y if SB is reduced to <3h/day (4) whereas prospective associations exist between SB with mortality and morbidity (2, 3). Short term experimental studies indicate that physical inactivity affects energy balance and is considered conducive to weight gain (5, 6). A decrease in PA has a considerable ability to decrease total energy expenditure (TEE) without any compensatory changes in energy intake, which generate a positive energy balance. The extent to which reducing and breaking up SB over sustained periods of time considerably increases TEE has never been investigated under free-living conditions.

Our hypothesis are that, a daily 3h reduction of SB during 1-week, either by increasing the number of breaks and by shifting SB to low intensity physical activity (LIPA), mainly through standing and walking activities, would substantially increase physical activity energy expenditure (PAEE) in male and female overweight/obese inactive computer desk workers compared to 1-week of usual prolonged SB. Prior to intervention, number of steps/day and PA were assessed through the use of a pedometer and accelerometer to respectively identify the habitual daily steps and to assure participants are inactive (<30 min/day of MVPA and ~ 5000 steps/day). Eligible participants were enrolled in a crossover experiment with two conditions performed in a random order: intervention (3h-reduction in SB) and control (habitual SB), both under free-living conditions. Each condition last for 1 week and participants were instructed to keep the same eating patterns while wearing an accelerometer, pedometer, a combined accelerometer and heart rate device, and an inclinometer (activpal). Doubly labeled water (DLW) was administered in both conditions to assess TEE, indirect calorimetry was employed to measure resting energy expenditure (REE), and PAEE subtracted from the sum of REE and thermogenic effect of food (assumed as 10% of TEE). Body composition was assessed at baseline and in the last day of the intervention week with DXA and participants wore the devices 24 hours a day during the two weeks and did the food records in three days in each week. In practice, at the workplace, our intervention to reduce SB include a software that hourly alert the participants to break up SB for approximately 7 minutes through adopting walking behaviors (~30-60 minutes/day) while during transportation, home/domestic, and leisure time contexts, an individual goal for number of steps/day was set based on an expected step cadence for ambulatory activities (~90-120 minutes/day). Also a number of strategies to break up SB were transmitted to the participants in the several contexts for accomplishing their goals.

At the workplace, daily breaks were automatically generated and registered through the software. Daily adherence in breaking up SB was supervised using phone calls during the day as well as compliance with the individual steps/day goal, self-registered in a diary at the end of the day. During the control week, supervision was performed to assure that participants remained inactive with a similar SB and number of steps/day, as observed at baseline.

During the trial, a 3-day food intake record was collected and analyzed at each condition. We anticipate that by using objective measures of transitions from sitting to standing and stepping, we will provide important methodological information, as sedentary time comprises a large proportion of waking hours and small changes may go undetected using self-report SB. A unique aspect of the present study is the utilization of state of-the-art technologies to investigate differences in daily EE and activity patterns in overweight/obese individuals.

The results of this project may have remarkable public health relevance. Most of the population weight gain in the past could have been avoided if a negative energy balance of 100 Kcal/day was achieved. We expect that our findings reveal a meaningful difference in energy expenditure by breaking up SB. We anticipated a public health message emphasizing "standing and walking more" as a simple approach to prevent weight gain and the rise of obesity in developed countries. This project may also contribute to disclose innovative energy balance -based methodologies for designing long-term intervention studies examining the effect of breaking up sedentary time on health-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participants were required to be sedentary, between 18-65 years old, have a BMI above 25.0 kg/m2 and physical inactive (not meeting the MVPA recommendations and not exceed 6000 steps/day). In addition subjects had to be free of any major disease with a general healthy status warranted.

Exclusion Criteria:

* Taking any medication or dietary supplements that may interfere with body composition or energy expenditure regulation, performing more than 5000 steps/day and meeting actual MVPA recommendations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from control week and intervention week in total energy expenditure (TEE) | week 1 and week 2
  The TEE was estimated by the doubly labeled water technique
Resting energy expenditure (REE) | Baseline (day 0)
  REE was measured by indirect calorimetry
Change from control week and intervention week in physical activity energy expenditure (PAEE) | week 1 and week 2
  PAEE was calculated as the difference between TEE and the sum of the REE and the thermogenic effect of food (assumed to be 10% of TEE)
Change from control week and intervention week in daily time spent in sedentary (SB) | week 1 and week 2
  PA variables were assessed using an accelerometer, a combined device that measures accelerometry and heart rate (actiheart)
Change from control week and intervention week in light (LIPA), moderate and vigorous (MVPA) intensity activities | week 1 and week 2
  PA variables were assessed using an accelerometer, a combined device that measures accelerometry and heart rate (actiheart)
Change from control week and intervention week in number of breaks in sedentary time (BST) | week 1 and week 2
  PA variables were assessed using an accelerometer, a combined device that measures accelerometry and heart rate (actiheart), and an inclinometer (activpal)
Change from control week and intervention week in time spent sitting (TSS) | week 1 and week 2
  An inclinometer (activpal)
Change from control week and intervention week in time spent standing (TSst) | week 1 and week 2
  An inclinometer (activpal)
Change from control week and intervention week in time spent walking (TSW) | week 1 and week 2
  An inclinometer (activpal)
Change from control week and intervention week in number of steps | week 1 and week 2
  Steps were assessed using an accelerometer, a combined device that measures accelerometry and heart rate (actiheart), an inclinometer (activpal) and a pedometer.

SECONDARY OUTCOMES:
Change from baseline and intervention week in body composition | Baseline (day 0) and final day of intervention week
  Body composition was assessed by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Analiza M Silva, PhD, Principal Investigator — Faculty of Human Kinetics, University of Lisboa
Locations (1):
- Exercise and Health Laboratory, Faculty of Human Kinetics, University of Lisboa, Cruz Quebrada, Lisbon District, Portugal

REFERENCES:
- [Derived] Judice PB, Teixeira L, Silva AM, Sardinha LB. Accuracy of Actigraph inclinometer to classify free-living postures and motion in adults with overweight and obesity. J Sports Sci. 2019 Aug;37(15):1708-1716. doi: 10.1080/02640414.2019.1586281. Epub 2019 Mar 7. PMID 30843462
- [Derived] Judice PB, Hamilton MT, Sardinha LB, Silva AM. Randomized controlled pilot of an intervention to reduce and break-up overweight/obese adults' overall sitting-time. Trials. 2015 Nov 2;16:490. doi: 10.1186/s13063-015-1015-4. PMID 26525049
- [Derived] Judice PB, Santos DA, Hamilton MT, Sardinha LB, Silva AM. Validity of GT3X and Actiheart to estimate sedentary time and breaks using ActivPAL as the reference in free-living conditions. Gait Posture. 2015 May;41(4):917-22. doi: 10.1016/j.gaitpost.2015.03.326. Epub 2015 Mar 30. PMID 25852024